CLINICAL TRIAL: NCT02655250
Title: The Neonatal Microbiome Study: Validity of Biologic Sample Collection Methods
Brief Title: Neonatal Microbiome Validity Study
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Amy E. Millen, Principal Investigator, State University of New York at Buffalo
Other Study IDs: 758632-1
Record Dates: First submitted 2015-06-19; First posted 2016-01-14 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Gut Microbiome
MeSH Terms: interventions — Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool and breast milk samples will be collected. Bacterial DNA will be isolated and stored. Human DNA will not be retained in these samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Microbiome

SUMMARY:
This is a validation study to compare proposed field collection methods with a gold standard collection technique for microbiome analysis of stool and breast milk samples.

DETAILED DESCRIPTION:
In order to conduct a future study of the gut microbiome in a population living in a rural, low income setting, this validation study will be conducted to verify the validity of our proposed field collection methods for stool and breast milk samples. We will compare the microbial diversity and abundance in the biologic samples using various proposed field collection methods to an immediately frozen sample. The proposed field collection methods are feasible for use in a community-based study in a low income setting with limited access to cold storage.

ELIGIBILITY:
Inclusion Criteria:

* Lactating women (for breast milk sample)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A convenience sample of men/women willing to provide a stool sample and/or breast milk sample.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Difference in intestinal microbiome between gold standard and proposed field protocol | Baseline
  Comparison of microbiome from snap-frozen sample (gold standard) to proposed field collection methods to determine which field method best correlates with the snap-frozen sample.
Difference in breast milk microbiome between gold standard and proposed field protocol | Baseline
  Comparison of microbiome from snap-frozen sample to proposed field collection methods to determine which field method best correlates with the snap-frozen sample.

CONTACTS AND LOCATIONS:
Overall Officials: Amy E Millen, PhD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- State University of New York at Buffalo, Farber Hall, Buffalo, New York, United States